CLINICAL TRIAL: NCT01050972
Title: Effectiveness of a Cognitive and Physical Intervention to Reduce Head and Muscle Pain in a Population of an Extensive Territory
Brief Title: Effectiveness of a Cognitive and Physical Intervention to Reduce Head and Muscle Pain in a Large Population
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: Fondazione CRT, Torino (Unknown); Turin, Italy (Other); Regione Piemonte (Other)
Responsible Party: Franco Mongini/ Professor and chairman, Unit of Headache and Facial Pain, Dept. of Clinical Pathophysiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Migraine; Tension Type Headache; Cervical Pain
Keywords: Headache; Cervical Pain; Cognitive treatment; Relaxation; Exercise
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Neck Pain; Headache; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive and physical program (Experimental): Experimental: Cognitive and physical program. Non randomized residents in the territory of Piedmont (Piemonte) Italy.
  Interventions: Behavioral: Behavioral: Cognitive, Relaxation, Exercise Therapy

INTERVENTIONS:
Behavioral: Behavioral: Cognitive, Relaxation, Exercise Therapy — Behavioral: Cognitive, Relaxation, Exercise Therapy The intervention consists of brief shoulder and neck exercises to be performed several times a day, a relaxation exercise and instructions of how to reduce hyperfunction of the craniofacial and cervical muscles during the day

SUMMARY:
This study is an interventional trial to evaluate the effectiveness of a cognitive and physical program (Intervention), in reducing the frequency of head and neck pain in the population of an extensive territory of Italy.

DETAILED DESCRIPTION:
In a previous non-randomized-controlled study in which the cognitive and physical programme was applied to a consistent number of office workers, a significant reduction of frequency of pain in the head and neck areas and of analgesic drug consumption was obtained. The results were stable at a 12 month follow up. More recently a controlled, cluster randomised, interventional trial was conducted on 1930 local government employees of the Municipality of Turin. The data obtained confirm those of the previous studies.

The present study was designed to confirm the data in a much more extensive population , that is, residents of the Italian Region Piemonte (Piedmont) who will apply to participate.

Primary objective is to confirm the effectiveness of the cognitive and physical programme (Intervention), in reducing the frequency of pain involving the head and neck area in a large population of a territory.

Secondary objective is to confirm the effectiveness of the Intervention, in reducing analgesic drugs consumption after the Intervention in the same population.

ELIGIBILITY:
Inclusion Criteria:

* All residents of the Region Piemonte (Italy) may apply for recruitment

Exclusion Criteria:

* Because of the pragmatic design, no exclusion criteria are required for this study

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in number of days per month with headache and shoulders pain after 12 months. | 24 months

SECONDARY OUTCOMES:
Reduction in number of days per month of drug intake after 12 months | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Franco Mongini, MD, Prof., Principal Investigator — Headache and Facial Pain Unit Dept. Clinical Pathophysiology University of Turin
Locations (1):
- Headache and Facial Pain Unit University of Turin, Turin, Italy